CLINICAL TRIAL: NCT04649424
Title: Comparative Evaluation of Nasopharyngeal Swabs for Sampling and Detection of SARS-CoV2
Brief Title: COVID-19 Nasal Swab Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Innovation Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B2020:121
Record Dates: First submitted 2020-11-27; First posted 2020-12-02 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CanSwab - 1st (Experimental): CanSwab will be swabbed first
  Interventions: Device: CanSwab
- CanSwab - 2nd (Experimental): CanSwab will be swabbed second.
  Interventions: Device: CanSwab

INTERVENTIONS:
Device: CanSwab — New nasopharyngeal swab design.

SUMMARY:
The purpose of this trial is to compare 2 types of nasonasopharyngeal swabs (a new design to a conventional nylon-flocked nasopharyngeal swab) for effectiveness.

DETAILED DESCRIPTION:
Compare the Precision ADM "CanSwab" nasopharyngeal swab to a conventional nylon-flocked nasopharyngeal swab on the basis of:

1. The amount of SARS-CoV2 virus (COVID-19) collected by swabs, measured in CT (thermal cycles)
2. Clinical concordance rate
3. Patient comfort during nasopharyngeal sampling procedure

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Ability to provide informed consent
* COVID-19 positive cohort only: a previous, positive COVID-19 test in the last 5 days and patient remains symptomatic

Exclusion criteria:

* Malformation of the base of the known skull
* Active nosebleed before the start of the sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Amount of SARS-CoV2 virus (COVID-19) collected | Baseline
  amount of SARS-CoV2 virus (COVID-19) collected measured in CT (thermal cycles).
Clinical concordance rate | Baseline
  Calculate approximate sensitivity and specificity of the CanSwab to the Flocked swab control.
Patient comfort | Baseline
  Patient description of comfort level between the 2 swabs experience measured by "Worse", "Identical" or "Better"

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — Health Sciences Centre
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No